CLINICAL TRIAL: NCT00100867
Title: Assessment of Safety and Toxicity Among Infants Born to HIV-1-Infected Women Enrolled in Antiretroviral Treatment Protocols in Diverse Areas of the World
Brief Title: Effects of Maternal Anti-HIV Treatment on Infants Born to HIV-Infected Women
Status: Completed | Type: Observational
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACTG A5190-P1054; 1U01AI068636 (NIH)
Record Dates: First submitted 2005-01-06; First posted 2005-01-07 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: HIV Infections
Keywords: Perinatal Transmission; Mother-to-Child Transmission
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine collection

SUMMARY:
In clinical trials being conducted throughout the world, pregnant HIV-infected women are given anti-HIV drugs before, during, and after they give birth to prevent mother-to-child transmission of HIV. However, the effects of this anti-HIV treatment on infants is unknown. The purpose of this study is to determine the safety, toxicity, and potential side effects of maternal anti-HIV treatment on infants born to these HIV-infected women.

Study hypothesis: Specific combination antiretroviral regimens used in clinical trials in diverse areas of the world are safe and well tolerated during pregnancy and breastfeeding periods, and are not associated with adverse side effects to the fetus, neonate, and/or breastfeeding infant. These regimens are associated with reduction of mother-to-child HIV transmission.

DETAILED DESCRIPTION:
Many HIV-infected women outside the United States enroll in clinical trials that provide them antiretroviral therapy (ART) to prevent mother-to-child transmission of HIV. However, data are limited on the safety, toxicity, and adverse effects that maternal ART may have on infants born to HIV-infected women. This study will monitor the adverse effects and potential benefits of maternal ART on these infants.

No antiretrovirals will be given in this study. This study will last 18 months. Infants will be enrolled in the study within 48 hours of birth. There will be 6 study visits starting at study entry and every 6 weeks thereafter. Infants will undergo blood and urine collection, and medical history assessments will occur at every visit. Mothers will also be evaluated at these visits.

ELIGIBILITY:
Inclusion Criteria:

* Infant born to HIV-1 infected mother enrolled in NIH-sponsored, international antiretroviral treatment trial AND who has had either in utero or postpartum antiretroviral exposure
* Parent or guardian willing to provide informed consent

Exclusion Criteria:

* Infant with no exposure to antiretrovirals OR who received only intrapartum antiretroviral exposure

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Infants born to HIV-infected women
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2006-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Nielsen, MD, MPH, Study Chair — University of California, Los Angeles; Judith S. Currier, MD, MSc, Study Chair — Center for AIDS Research and Education, University of California, Los Angeles
Locations (23):
- Botswana (2):
  - The Gaborone BHP Study Clinic, Gaborone
  - The Molepolole BHP Study Clinic, Gaborone
- Brazil (3):
  - Instituto de Pesquisa Clinica Evandro Chagas Fiocruz, Fundacao Oswaldo Cruz, Rio de Janeiro
  - Hospital dos Servidores do Estado, Rio de Janeiro
  - Hospital Geral de Nova Iguacu, Rio de Janeiro
- India (4):
  - YRG Center for AIDS Research and Education, Chennai
  - NARI AIDS Research Institute, Department of Clinical Science, Pune
  - NARI AIDS Research Institute, Dr. Kotnis Dispensary, Pune
  - NARI-NIV Clinic, Pune
- Malawi (2):
  - Univ. of Malawi, John Hopkins Project, Blantyre
  - University of North Carolina Project (UNC Project), Lilongwe
- Peru (2):
  - Asociacion Civil IMPACTA Salud y Educacion,, Miraflores, Lima region
  - Asociacion Civil IMPACTA Salud y Educacion, Lince, Lima
- South Africa (2):
  - Perinatal HIV Research Unit at Chris Baragwanath Hospital, Johannesburg
  - University of the Witwatersrand, Johannesburg
- Thailand (7):
  - Siriraj Hospital, Bangkok Noi, Bankok
  - Chonburi Regional Hospital, Chonburi, Muang, Changwat Chon Buri
  - Phayao Provincial Hospital, Phayao, Tambol Mae Sai, Muang Phayao
  - Bhumibol Adulyadej Hospital, Bangkok, Bangkok
  - Chiang Mai University, Chang Mai
  - Institut de Recherche pour Developpement (IRD), Chiang Mai
  - Prapokklao Hospital Chantaburi, Muang Chantaburi
- University of Zimbabwe, Harare, Zimbabwe

REFERENCES:
- [Background] Abrams EJ. Prevention of mother-to-child transmission of HIV--successes, controversies and critical questions. AIDS Rev. 2004 Jul-Sep;6(3):131-43. PMID 15595430
- [Background] Scarlatti G. Mother-to-child transmission of HIV-1: advances and controversies of the twentieth centuries. AIDS Rev. 2004 Apr-Jun;6(2):67-78. PMID 15332429
- [Background] Semprini AE, Fiore S. HIV and pregnancy: is the outlook for mother and baby transformed? Curr Opin Obstet Gynecol. 2004 Dec;16(6):471-5. doi: 10.1097/00001703-200412000-00006. PMID 15534442
- [Background] Sullivan JL. Prevention of mother-to-child transmission of HIV--what next? J Acquir Immune Defic Syndr. 2003 Sep;34 Suppl 1:S67-72. doi: 10.1097/00126334-200309011-00010. PMID 14562860